CLINICAL TRIAL: NCT01322724
Title: Comparing Warm Versus Cool Temperature Water During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 00007299
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Colonoscopy
Keywords: colonoscopy; colon cancer screening; patient discomfort scores; sedation medication requirements; water insertion method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warm water (Active Comparator): Body temperature (95-100 degrees F) water
  Interventions: Procedure: Warm vs Cool water
- Cool water (Experimental): Room temperature (68-73 degrees F) water
  Interventions: Procedure: Warm vs Cool water

INTERVENTIONS:
Procedure: Warm vs Cool water — Body vs Room temperature water used during insertion of colonoscopy

SUMMARY:
The purpose of this study will be to determine if the temperature of water used during insertion of colonoscopy makes a difference in patient discomfort and sedation requirements. The hypothesis of this study is patients receiving screening colonoscopy utilizing the water insertion method with room temperature (cool) water will have similar pain scores and medication requirements compared to water insertion method using body temperature (warm) water.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 85 years undergoing elective outpatient screening colonoscopy for colon cancer screening

Exclusion Criteria:

* Patients undergoing colonoscopy for any other indication besides colon cancer screening
* Patients with prior colonic resections
* Patients with chronic narcotic or benzodiazepine use
* Poor bowel preparation (i.e. Boston bowel preparation score < 8)
* Patients with obstructing colonic lesions detected on colonoscopy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dose of sedation medication used (fentanyl and midazolam) | Duration of the colonoscopy; Up to 3 hours

SECONDARY OUTCOMES:
Patient pain/discomfort score | During the day of the procedure; Up to 1 day

CONTACTS AND LOCATIONS:
Overall Officials: M. Brian Fennerty, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Lee BY, Katon R, Herzig D, Fennerty MB. Warm water infusion during sedated colonoscopy does not decrease amount of sedation medication used. Gastrointest Endosc. 2012 Dec;76(6):1182-7. doi: 10.1016/j.gie.2012.08.002. Epub 2012 Sep 26. PMID 23021168